CLINICAL TRIAL: NCT07065409
Title: Phase I Clinical Trial of Induced Pluripotent Stem Cell-derived Extracellular Vesicles Combined With Temporal Muscle Flap Application in Promoting Intracranial and Extracranial Blood Flow Reconstruction in Patients With Moyamoya Disease
Brief Title: Treatment of Moyamoya Disease With iPSC-derived Exosomes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huaqiu Zhang (Other)
Responsible Party: Sponsor-Investigator, Huaqiu Zhang, Clinical Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202503034
Record Dates: First submitted 2025-05-09; First posted 2025-07-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Moyamoya Disease
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPSC-EVs (Experimental)
  Interventions: Biological: iPSC-EVs

INTERVENTIONS:
Biological: iPSC-EVs — iPSC-EVs，The drug number is NouvSoma002-01. It is from iRegene Therapeutics Co., Ltd.

SUMMARY:
Moyamoya disease is a cerebrovascular disease clinically characterized by chronic progressive stenosis or occlusion at the ends of bilateral internal carotid arteries and the origin of anterior cerebral arteries and middle cerebral arteries, followed by the formation of abnormal vascular networks at the base of the skull. Clinically, patients with Moyamoya disease mainly present with ischemic or hemorrhagic stroke, and there are two peaks of incidence in children aged 3-5 and middle-aged people aged 40-50. Moreover, as the pathogenesis and treatment evaluation of Moyamoya disease are still in the research trough at present, new discoveries are prone to occur and thus attract a great deal of attention. It not only has a beneficial promoting effect on the treatment and diagnosis of patients, but also makes it easier for research topics to be reported in top journals.

This study intends to combine iPSC-EVs local skin transplantation with temporal muscle application to promote muscle angiogenesis and the establishment of extracranial and intracranial collateral circulation after temporal muscle application. The above-mentioned design features high efficiency, safety and convenience, and is an innovative exploration both at home and abroad. We hope to screen out safe, efficient and simple preparation methods and transplantation methods of iPSC-EVs through systematic experiments, establish an effective clinical evaluation system, and provide auxiliary means for intracranial and extracranial blood flow reconstruction surgery in the treatment of Moyamoya disease. Moreover, in terms of topic selection, iPSC is currently one of the most promising directions for innovative treatment worldwide.

DETAILED DESCRIPTION:
Moyamoya disease is a cerebrovascular disease clinically characterized by chronic progressive stenosis or occlusion at the ends of bilateral internal carotid arteries and the origin of anterior cerebral arteries and middle cerebral arteries, followed by the formation of abnormal vascular networks at the base of the skull. Because this abnormal vascular network at the base of the skull looks like wisps of smoke on cerebral angiography, the Japanese Suzuki first named it "Moyamoya Disease" in the 1960s. Clinically, patients with Moyamoya disease mainly present with ischemic or hemorrhagic stroke, and there are two peaks of incidence in children aged 3-5 and middle-aged people aged 40-50. Epidemiological studies have found that Moyamoya disease is mainly distributed among the population in East Asia, including Japan, South Korea and China, and its incidence rate in China has shown a significant upward trend in recent years.Moreover, as the pathogenesis and treatment evaluation of Moyamoya disease are still in the research trough at present, new discoveries are prone to occur and thus attract a great deal of attention. It not only has a beneficial promoting effect on the treatment and diagnosis of patients, but also makes it easier for research topics to be reported in top journals.

In recent years, with the popularity of IPscs, the emerging therapeutic approach of extracellular vesicles derived from IPscs (iPSC-EVs) has gradually come into the public view. Extracellular vesicles derived from IPscs have specific bioactive substances related to iPSC functions. Their main advantages are manifested as follows: (1) They have a strong ability to promote regeneration and can promote vascular regeneration; (2) It has a powerful function of inhibiting inflammatory responses and can significantly inhibit the release of inflammatory factors by microglia, astrocytes and oligodendrocytes. (3) The homogeneity and stability of IPscs enable extracellular vesicles derived from IPscs to have high drugability; (4) IPscs have good potential for gene editing and can support the engineering of extracellular vesicles and drug delivery in extracellular vesicles. (5) The homing effect of IPSC-differentiated cells can endow the corresponding extracellular vesicles with better tissue-targeting characteristics.

This study intends to combine iPSC-EVs local skin transplantation with temporal muscle application to promote muscle angiogenesis and the establishment of extracranial and intracranial collateral circulation after temporal muscle application. The above-mentioned design features high efficiency, safety and convenience, and is an innovative exploration both at home and abroad. We hope to screen out safe, efficient and simple preparation methods and transplantation methods of iPSC-EVs through systematic experiments, establish an effective clinical evaluation system, and provide auxiliary means for intracranial and extracranial blood flow reconstruction surgery in the treatment of Moyamoya disease. Moreover, in terms of topic selection, iPSC is currently one of the most promising directions for innovative treatment worldwide.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed adult patients with MMD aged 18-75 years (inclusive), with bilateral terminal occlusion of the internal carotid arteries (ICA) and stenosis or occlusion of the anterior cerebral artery (ACA) and middle cerebral artery (MCA) at the origin, accompanied by the formation of abnormal vascular networks at the base of the skull, as indicated by head DSA or MRA. Unilateral or bilateral lesions are acceptable. Suzuki score ≥ 3.
2. Relevant bone marrow, liver, kidney, and heart function indicators meet the following standards (based on the normal values of the clinical trial center): absolute neutrophil count (ANC) ≥ 1.5×109/L, platelets ≥ 100×109/L, total serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), ALT, AST, or ALP ≤ 3 times ULN; serum creatinine ≤ 1.5 times ULN, international normalized ratio (INR) ≤ 1.5 times ULN, APTT ≤ 1.5 times ULN.
3. Patients have undergone temporal muscle patch surgery and have not achieved satisfactory improvement in symptoms.
4. Patients have been followed up for ≥ 3 months since the surgery.
5. Vascular DSA performed 3 months after the surgery indicates poor blood flow reconstruction.
6. CTP or ASL performed 3 months after the surgery shows ischemia.
7. Patients still have clinical manifestations of cerebral ischemia or cerebral infarction due to MMD 3 months after the surgery.
8. Patients or their legal representatives have given informed consent and signed the informed consent form.

Exclusion criteria:

1. Patients with severe liver or kidney dysfunction or other complications;
2. Patients with a history of mental disorders or mental diseases;
3. Patients with coagulation disorders;
4. Patients with extensive cerebral infarction or in a coma;
5. Patients who only undergo direct bypass surgery;
6. Patients who have not signed the surgical consent form;
7. Patients with allergic constitutions or a clear history of allergies;
8. Pregnant women, lactating women, and patients with plans to conceive during the trial period;
9. Patients who have participated in other clinical trials in the past three months;
10. Patients deemed unsuitable for the trial by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 Day、2 week、1 month
  Evaluate the tolerance and adverse reactions of patients after 3 days, 2 weeks and 1 month of iPSC-EVs treatment.
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability].
Imaging examinations | 1 month
  Imaging examinations were conducted on the patients before iPSC-EVs treatment, and at 1 month after treatment.
  Imaging examinations: MRI and TCD.
Neuropsychological tests | 1 month
  Neuropsychological tests were conducted on the patients before iPSC-EVs treatment, and at 1 month after treatment.
  neuropsychological tests: mRS, MMSE and MoCA

SECONDARY OUTCOMES:
Imaging examinations | 3 month, 6 month, 12 month, and 24 month
  Imaging examinations for post-treatment imaging assessment of blood flow reconstruction function.
  Imaging examinations: DSA, MRI, CTP, TCD, HR-VWI, and CT.
Neuropsychological tests | 3 month, 6 month, 12 month, and 24 month
  Neuropsychological tests for post-treatment imaging assessment of blood flow reconstruction function.
  neuropsychological tests: mRS, MMSE and MoCA

CONTACTS AND LOCATIONS:
Overall Officials: Huaqiu Zhang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No